CLINICAL TRIAL: NCT02881489
Title: Evaluation of Mesenchymal Stem Cell Culturing Protocols in the Treatment of Amyotrophic Lateral Sclerosis
Brief Title: Autologous Bone Marrow Mesenchymal Stem Cells in the Treatment of Patients With Amyotrophic Lateral Sclerosis
Acronym: UwmBmmscALS
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Warmia and Mazury (Other)
Responsible Party: Principal Investigator, Wojciech Maksymowicz, MD, PhD, Professor, University of Warmia and Mazury
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UWM/ALS-MSC.2015/002
Record Dates: First submitted 2016-04-22; First posted 2016-08-29 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2016-08

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Autologous BM-MSCs injection (Experimental): Intervention: Biological: Cell-based therapy of autologous bone marrow-derived mesenchymal stem cells which are transplanted intrathecally (via a standard lumbar puncture) into the ALS subjects.
  Interventions: Other: Biological: Cell-based therapy

INTERVENTIONS:
Other: Biological: Cell-based therapy — Human autologous bone marrow-derived mesenchymal stem cell transplantation in ALS patients.

SUMMARY:
The goal of this study is to investigate the safety and tolerability of autologous bone marrow-derived mesenchymal stem cells administration in the individuals with diagnosed amyotrophic lateral sclerosis.

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis (ALS) is one of the progressive neurodegenerative disorders, affecting upper and lower motor neurons in the cerebral cortex, brainstem and spinal cord. Hence, the signs of damage motor neurons are both at the peripheral (eg. atrophy), and central (eg. spasticity) level. There is no effective treatment for ALS and the majority of patients die within 5 years after diagnosis, usually due to respiratory failure. Numerous studies on murine models revealed that mesenchymal stem cells (MSCs) successfully improve the clinical and pathological features of ALS. The goal of this nonrandomized, open label study is to investigate the safety and tolerability of autologous bone marrow-derived mesenchymal stem cell transplantation into the individuals with diagnosed amyotrophic lateral sclerosis. This clinical trial is conducted to test the therapeutic (neuroprotective and paracrine) effect of autologous bone marrow-derived mesenchymal stem cells (BM-MSCs). All patients enrolled will have a documented history of ALS disease prior to study enrollment. Patients are recruited for a clinical trial not longer than 1 year from disease diagnosis. Then, patients are divided into two groups: Group I - patients receiving intrathecally one application of BM-MSCs and Group II - patients receiving intrathecally three applications (each administration every two months) of BM-MSCs. Subsequently, autologous bone marrow-derived mesenchymal stem cell transplantation to the cerebrospinal fluid at the site of the spinal cord will be performed. Finally, treatment safety, adverse events and exploratory parameters, including electromyographic (EMG) studies, forced vital capacity (FVC) and functional rating scale (FRS) to establish ALS progression rate will be recorded throughout the duration and in the post-treatment follow up period.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of the ALS disease before the cell transplantation (diagnose established following the El Escorial criteria for definite ALS)
* good understanding of the protocol and willingness to consent
* signed informed consent
* disease duration: up to 2 years
* FVC > 50% / pulmonologist certificate about respiratory function of the patient

Exclusion Criteria:

* cancer,
* autoimmune diseases
* renal failure,
* subject is a respiratory dependent.
* subject unwilling or unable to comply with the requirements of the protocol
* pregnancy, breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-11; Primary Completion 2018-04 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Changes in the Amyotrophic Lateral Sclerosis Functional Rating Scale (ALSFRS) between patients before and after stem cell transplantation. | From day of enrolment until the date of first stem cell injection (6 months - first time ALSFRS) + and then every 2 months up to 1,5 year of the trial
  ALSFRS is ordinal rating scale questionnaire (rating 0-4 for each question, 4 is most functional, 0-48 total) of 12 functional activities. The most functional total score is 48. The First time the ALSFRS questionnaire has been dane after enrolment of the patients and then after 6 months of observation and stem cell injections the ALSFRS has been dane every 2 months up to 1,5 year of follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Wojciech Maksymowicz, MD, Prof., Principal Investigator — Faculty of Medical Sciences, University of Warmia and Mazury in Olsztyn, Poland

IPD SHARING:
Plan to Share IPD: Undecided